CLINICAL TRIAL: NCT00514137
Title: A Phase II Trial of Sunitinib (SU11248) in Multiple Myeloma
Brief Title: Sunitinib in Treating Patients With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00208; MC058F; CDR0000560703 (Registry Identifier: PDQ (Physician Data Query)); N01CM62205 (NIH)
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-03

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (kinase inhibitor therapy) (Experimental): Patients receive 37.5 mg oral sunitinib malate once daily on days 1-42. Treatment repeats every 42 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Oral 37.5 mg each day of the 6-week cycle (continuous dosing).
  Other Names: SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial is studying how well sunitinib works in treating patients with relapsed multiple myeloma. Sunitinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the number of responses in patients with relapsed multiple myeloma treated with sunitinib (sunitinib malate).

SECONDARY OBJECTIVES:

I. To assess the toxicity of sunitinib malate in patients with relapsed multiple myeloma.

II. To assess time to progression after initial response to sunitinib malate.

OUTLINE:

Patients receive oral sunitinib malate once daily on days 1-42. Treatment repeats every 42 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed multiple myeloma
* Measurable disease as defined by at least one of the following:

  * Serum monoclonal protein ≥ 1.0 g by protein electrophoresis
  * Urine monoclonal protein > 200 mg by 24-hour electrophoresis
  * Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis ≥ 30%
* Not a candidate for stem cell transplantation OR have undergone prior stem cell collection
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,000/microliter (mcL)
* Platelets ≥ 75,000/mcL
* Hemoglobin ≥ 8 g/dL
* Total serum bilirubin normal
* aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal
* Creatinine < 2.5 mg/dL
* Negative pregnancy test for women of childbearing potential
* No more than 4 prior therapies

  * Stem cell transplantation and preceding induction therapy will be considered 1 therapy
* Prior anthracycline exposure or central thoracic radiotherapy that included the heart in the radiotherapy port allowed provided patient has a New York Heart Association (NYHA) class II or better cardiac function on baseline ECHO or multiple gated acquisition scan (MUGA)
* Concurrent bisphosphonates allowed
* At least 7 days since prior and no concurrent cytochrome P450 3A4 (CYP3A4) inhibitors
* At least 12 days since prior and no concurrent CYP3A4 inducers

Exclusion Criteria:

* Pregnant or nursing women
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib malate
* History of serious ventricular arrhythmia or corrected QT interval (QTc) prolongation
* Poorly controlled hypertension
* Any condition that impairs the ability to swallow and retain sunitinib malate tablets
* Patients with a preexisting thyroid abnormality who are unable to maintain thyroid function in the normal range with medication
* Other active malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix or breast
* Concurrent uncontrolled illness including, but not limited to, ongoing or active infections or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who have not recovered from adverse events of prior therapy
* Chemotherapy or radiotherapy ≤ 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study entry
* Any major surgery ≤ 4 weeks prior to study entry
* Nonmyelosuppressive agents ≤ 2 weeks prior to study entry
* Any other prior antiangiogenic agents
* Concurrent high-dose corticosteroids

  * Concurrent chronic steroids (up to 20 mg/day prednisone equivalent) allowed for disorders other than amyloid; NOTE: Bisphosphonates are considered to be supportive care rather than therapy, and are thus allowed while on protocol treatment
* Concurrent therapeutic doses of coumarin-derivative anticoagulants
* Concurrent agents with proarrhythmic potential
* Concurrent combination antiretroviral therapy for HIV-positive patients
* Any other concurrent investigational agents or anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Research Consortium, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen participants were accrued from September 2007 to December 2008.
Pre-assignment Details: All 13 participants were analyzed.
Groups:
- Treatment (Kinase Inhibitor Therapy): Patients receive oral sunitinib malate once daily on days 1-42. Treatment repeats every 42 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 61 [53 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 11
  Hong Kong | 1
  Singapore | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Confirmed Responses (Complete Response [CR], Very Good Partial Response [VGPR], or Partial Response [PR])
Description: A confirmed response is defined as a patient who has achieved response and maintained it on two consecutive evaluations at least 2 weeks apart.
  A Complete Response (CR) is defined as the complete disappearance of an M-protein and fewer than 5% bone marrow plasmacytosis.
  A Hematologic Very good partial response (VGPR) is defined as having a ≥ 90% reduction of M-protein from serum, a Urine M-spike to be ≤ 100 mg/24 hours, and a disappearance of soft tissue plasmacytomas.
  A Partial Response (PR) is defined as having a 50-89% reduction in the level of the serum monoclonal protein, a reduction in 24-hour urinary light chain excretion either by ≥90% or to <200 mg, and a ≥ 50% reduction in size of soft tissue plasmacytoma.
Time Frame: Every 6 weeks from the first initiation of therapy up to 72 weeks
Population: All 13 participants were evaluable for a response
Measure: Number; unit: participants
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 13
participants | 0

2. Secondary Outcome: Event-free Survival
Description: The distribution of progression-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to progression or death due to any cause, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 13
months | 2.86 [1.35 to 5.52]

3. Secondary Outcome: Duration of Response
Description: The distribution of duration of response will be estimated using the method of Kaplan-Meier.
Time Frame: From the documentation of response until the date of progression
Population: No analysis was done because there were no confirmed responses.
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Toxicity
Description: Assessed per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Included are the toxicities at least possibly related to the study drug.
Time Frame: From the time of first treatment to up to 30 days after the last day of study drug treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Number analyzed (Participants) | 13
participants
  Grade 3+ Adverse Events | 10
  Grade 4+ Adverse Events | 3
  Grade 5 Adverse Events | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Kinase Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Kinase Inhibitor Therapy) (N=13)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Kinase Inhibitor Therapy) (N=13)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (9)
Hypothyroidism (Endocrine disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 4 (6)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 5 (6)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 11 (19)
Fever (General disorders) | 2 (2)
Amylase increased (Investigations) | 2 (3)
Leukocyte count decreased (Investigations) | 9 (11)
Lipase increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 7 (10)
Platelet count decreased (Investigations) | 10 (14)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 5 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (5)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (3)
Hypertension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less